CLINICAL TRIAL: NCT02318797
Title: Optimizing Behavioral Health Homes by Focusing on Outcomes That Matter Most for Adults With Serious Mental Illness
Brief Title: Optimizing Behavioral Health Homes for Adults With Serious Mental Illness
Acronym: PCORI OH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: UPMC Center for High-Value Health Care (Unknown); Western Psychiatric Institute and Clinic of UPMC (Unknown); Community Care Behavioral Health Organization (Unknown); Columbia Montour Snyder Union Mental Health (Unknown); Behavioral Health Alliance of Rural Pennsylvania (Unknown)
Responsible Party: Principal Investigator, Charles Reynolds, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PCORI 271
Record Dates: First submitted 2014-11-25; First posted 2014-12-17 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Chronic Disease; Mental Health; Behavioral Health; Cardiovascular Disease; Diabetes Mellitus Type 2; Substance-related Disorders; Vascular Diseases
Keywords: Chronic disease; Mental Health; Behavioral Health; Community mental health centers; Intervention studies; Mixed methods; Qualitative research
MeSH Terms: conditions — Chronic Disease; Psychological Well-Being; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Substance-Related Disorders; Vascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Self-Directed Care (Active Comparator): See intervention description
  Interventions: Behavioral: Patient Self-Directed Care
- Provider-Supported Integrated Care (Active Comparator): See intervention description
  Interventions: Behavioral: Provider-Supported Integrated Care

INTERVENTIONS:
Behavioral: Patient Self-Directed Care — Patient self-management toolkits, web portal with information on health conditions, personal health care use data, health tracking tools and wellness programs
  Arms: Patient Self-Directed Care
Behavioral: Provider-Supported Integrated Care — Registered nurse on staff at community mental health centers with access to patient-level physical health information to: 1) work with patients on coordinating their care, 2) enhance communication between providers and payer, and 3) provide patient wellness support and education
  Arms: Provider-Supported Integrated Care

SUMMARY:
Adults with serious mental illness (SMI) frequently have unmet medical needs which place them at risk for adverse health outcomes. While there are proven ways to manage and/or prevent serious medical conditions common among this population, information is needed to understand their impact on outcomes that matter most for patients, particularly in community mental health centers (CMHCs) where most adults with SMI receive their care and rural areas where locating and receiving health care services can be challenging.

The investigators will test two promising ways for promoting the health, wellness, and recovery of adults with SMI. One way will help patients manage their health and health care through self-management strategies, including the use of a web portal, and peer support (patient self-directed care) and the other through interactions with nurses during clinic visits (provider-supported integrated care).

The investigators will compare the two interventions on three primary patient-centered outcomes (i.e. patient activation in care, health status, engagement in primary/specialty care). The investigators hypothesize that:

1. Patient self-directed care will result in improvement in patient activation.
2. Provider-supported integrated care will result in greater improvement in frequency in primary/specialty care visits.
3. Both interventions will result in significant improvements in the three primary outcomes.

The investigators will collect information from patients, caregivers, and clinic staff at different points in time during the study. Patients will be asked to complete questionnaires and additional data on their service use will be gathered. Some patients and providers will also be interviewed about their experiences with care. The investigators will examine these data to learn if, how, and why the new services improve outcomes over time. This information will help us understand patient and other stakeholder views about the services and, if appropriate, ensure their continued and/or expanded availability.

DETAILED DESCRIPTION:
The combination of high medical need with difficulty accessing quality medical care makes adults with serious mental illness (SMI) one of our nation's most medically vulnerable populations. While evidence-based interventions exist for managing and/or preventing high rates of chronic medical conditions in this population, information is needed to understand their impact on outcomes that matter most for patients, particularly in community mental health centers (CMHCs) where most adults with SMI receive their care and rural areas where availability of and access to health care services is limited.

Building on the work of a multi-stakeholder collaboration in rural Pennsylvania, the UPMC Center for High-Value Health Care and our patient, provider, and payer partners will evaluate two promising interventions-patient self-directed care and provider-supported integrated care-for promoting the health, wellness, and recovery of adults with SMI. We will address four questions that patients have identified as important to them:

1. Given my mental and physical conditions, what should I expect will happen to my overall health, wellness, and recovery when I engage in the new services offered by my CMHC?
2. If I choose to participate in these services, what are the potential advantages or disadvantages to me?
3. In what ways can I become more active in managing my own health and health care?
4. Which of the services that my CMHC could make available to me will impact outcomes that I care about and help me make the best decisions about my health and care? Our aims compare the effectiveness of the interventions on patient-centered outcomes and explore the moderating role of patient characteristics and the mediating role of engagement in the interventions. By demonstrating which interventions improve outcomes for whom under what circumstances, we will inform positive patient heath choices and key stakeholder decision making to support these choices, thereby advancing health system improvement efforts to avoid early mortality and comorbidity in this population.

We have enrolled 1,229 Medicaid-enrolled adults who have or are at risk for chronic medical conditions and receive care at rural and suburban CMHCs. Using a cluster randomized design with a mixed-methods approach, we randomly assigned 11 CMHCs to one of the two interventions. Quantitative (self-report, claims, process) and qualitative (interviews) data will be gathered across multiple time points from baseline through the end of the two-year intervention. Descriptive and multivariate analyses will be used to examine the impact of the interventions on outcomes over time and explore the roles of moderating and mediating variables. Qualitative results will be used to understand patient and other stakeholder perspectives and promote dissemination and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Serious mental illness (schizophrenia, bipolar disorder, major depression)
* Receive services at one of the 11 participating community mental health centers
* At least one claim for outpatient case management or peer specialist services

Exclusion criteria:

* Not willing to provide informed consent
* Assessed by clinicians as being too ill to be treated on an outpatient basis
* Unable to speak, read, or understand English at the minimum required level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1229 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Reynolds, MD, Principal Investigator — University of Pittsburgh; UPMC Center for High-Value Health Care; James M. Schuster, MD, MBA, Principal Investigator — Community Care Behavioral Health; UPMC Center for High-Value Health Care; Tracy A. Carney, AAS, Principal Investigator — Recovery Central Clubhouse, Columbia Montour Snyder Union Mental Health
Locations (1):
- Community Care Behavioral Health Organizations, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Still determining data sharing plan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Started (# of individuals enrolled in each study arm) | 516 | 713
Completed (# of individuals for whom we have at least one data element at the final data collection time point) | 428 | 611
Not Completed | 88 | 102
Not completed — Death | 3 | 6
Not completed — Lost to Follow-up | 85 | 96

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care | Total
Number analyzed (Participants) | 516 | 713 | 1229
Age, Continuous [Mean (Full Range); unit: years] | 42.37 [18 to 76] | 43.47 [19 to 72] | 43.01 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341 | 428 | 769
  Male | 175 | 285 | 460
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 514 | 709 | 1223
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 72 | 93
  White | 483 | 621 | 1104
  More than one race | 11 | 15 | 26
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Activation in Care (PAM, a 13-item Scale)
Description: Assessed using the PAM, a 13-item scale that renders a total activation score. This measure gauges the knowledge, skills, and confidence of patients essential to managing their own health and health care. It divides into progressively higher levels of activation: starting to take a role, building knowledge and confidences, taking action, and maintaining behaviors. The raw score scale for the PAM ranges from 13 to 52. The activation scale for the PAM ranges from 0 to 100. The lower values represent a poor outcome while higher values represent a better outcome.
Time Frame: Baseline and every 6 months over 2 year active intervention period
Population: Includes those who completed the measure at baseline and whose measure was able to be scored (ie. was not missing data which would have rendered it unusable in analysis)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 438 | 615
units on a scale
  Baseline | 56.99 (15.03) | 56.77 (14.59)
  6-month follow up: number analyzed (Participants) | 277 | 463
  6-month follow up | 56.84 (14.45) | 58.74 (14.90)
  12-month follow up: number analyzed (Participants) | 227 | 415
  12-month follow up | 58.36 (15.08) | 57.46 (14.89)
  18-month follow up: number analyzed (Participants) | 218 | 354
  18-month follow up | 58.90 (14.98) | 57.84 (15.11)
  24-month follow up: number analyzed (Participants) | 145 | 303
  24-month follow up | 57.04 (15.15) | 58.61 (15.64)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment by time interaction; Test type: Superiority; p = 0.0019, Mixed Models Analysis

2. Primary Outcome: Change in Health Status ( SF-12v2™): Physical Health Sub-scale
Description: Health status is measured using the SF-12v2™, a widely used and practical health survey tool consisting of 12 questions and two sub-scales for measuring physical and mental health status and symptom effects and functioning. The physical health component summary score is created using a weighted sum of all 12 items and then a scoring algorithm places negative weights on four of the health domains and positive weights on the other four health domains. Scores range from 0-100 and better physical health is indicated by a higher score.
Time Frame: Baseline and every 6 months over 2 year active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 511 | 705
units on a scale
  Baseline | 42.12 (11.47) | 42.47 (11.05)
  6-month follow up: number analyzed (Participants) | 334 | 547
  6-month follow up | 41.19 (11.44) | 42.26 (11.00)
  12-month follow up: number analyzed (Participants) | 274 | 480
  12-month follow up | 41.33 (10.78) | 41.19 (11.32)
  18-month follow up: number analyzed (Participants) | 263 | 422
  18-month follow up | 39.71 (11.80) | 41.28 (10.99)
  24-month follow up: number analyzed (Participants) | 187 | 384
  24-month follow up | 40.07 (12.16) | 41.96 (10.99)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.4103, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time from baseline (only conducted if treatment by time interaction test non-significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment by time interaction; Test type: Superiority; p = 0.4068, Mixed Models Analysis
Statistical Analysis 4: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment interaction (only calculated if gender by treatment by time non-significant); Test type: Superiority; p = 0.2656, Mixed Models Analysis

3. Primary Outcome: Change in Engagement in Primary/Specialty Care
Description: The frequency of primary/specialty care visits over two 12-month time periods.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: Study participants who were Medicaid eligible for 80% of the year prior to the data collection time point
Measure: Mean (Standard Deviation); unit: Frequency of visits in 12-month periods
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
Frequency of visits in 12-month periods
  Baseline | 9.87 (7.93) | 8.72 (6.69)
  12-month follow up: number analyzed (Participants) | 440 | 620
  12-month follow up | 11.33 (8.46) | 11.77 (7.93)
  24-month follow up: number analyzed (Participants) | 310 | 582
  24-month follow up | 11.05 (8.58) | 10.88 (7.90)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.4582, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time from baseline (only conducted if treatment by time interaction test non-significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment by time interaction; Test type: Superiority; p = 0.05, Mixed Models Analysis
Statistical Analysis 4: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment interaction (only calculated if gender by treatment by time non-significant); Test type: Superiority; p = 0.1792, Mixed Models Analysis

4. Primary Outcome: Change in Health Status ( SF-12v2™): Mental Health Sub-scale
Description: Health status is measured using the SF-12v2™, a widely used and practical health survey tool consisting of 12 questions and two sub-scales for measuring physical and mental health status and symptom effects and functioning. The mental health component summary score is created using a weighted sum of all 12 items and then a scoring algorithm places negative weights on four of the health domains and positive weights on the other four health domains (reverse of the weighting used for the physical health component summary score). Scores range from 0-100 and better mental health is indicated by a higher score.
Time Frame: Baseline and every 6 months during the active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 510 | 703
units on a scale
  Baseline | 36.59 (11.91) | 39.57 (12.13)
  6-month follow up: number analyzed (Participants) | 334 | 547
  6-month follow up | 37.79 (11.18) | 40.78 (12.02)
  12-month follow up: number analyzed (Participants) | 274 | 480
  12-month follow up | 39.42 (10.35) | 39.80 (11.48)
  18-month follow up: number analyzed (Participants) | 263 | 422
  18-month follow up | 38.52 (11.15) | 40.63 (11.40)
  24-month follow up: number analyzed (Participants) | 187 | 384
  24-month follow up | 39.63 (11.38) | 40.56 (11.92)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.2179, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time from baseline (only conducted if treatment by time interaction test non-significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment by time interaction; Test type: Superiority; p = 0.4797, Mixed Models Analysis
Statistical Analysis 4: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for gender by treatment interaction (only calculated if gender by treatment by time non-significant); Test type: Superiority; p = 0.0014, Mixed Models Analysis

5. Secondary Outcome: Change in Hope (Hope Scale)
Description: Assessed using the Hope Scale, an instrument designed to measure hope that has been previously used in health services research. Twelve items are rated on a four-point response scale ranging from "definitely false" to "definitely true" and summed to produce a total score. The hope scale ranges from 1 to 10, with 1 being no hope and 10 being filled with hope.
Time Frame: Baseline and every 6 months during the active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 510 | 710
Units on a scale
  Baseline | 6.24 (2.59) | 6.46 (2.62)
  6 month follow-up: number analyzed (Participants) | 336 | 544
  6 month follow-up | 6.24 (2.52) | 6.57 (2.60)
  12 month follow-up: number analyzed (Participants) | 278 | 476
  12 month follow-up | 6.47 (2.47) | 6.56 (2.64)
  18 month follow-up: number analyzed (Participants) | 264 | 427
  18 month follow-up | 6.31 (2.47) | 6.65 (2.53)
  24 month follow-up: number analyzed (Participants) | 188 | 380
  24 month follow-up | 6.35 (2.47) | 6.51 (2.61)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.0058, Mixed Models Analysis

6. Secondary Outcome: Change in Quality of Life (QLESQ)
Description: Patient quality of life is measured using the QLESQ (Quality of Life Enjoyment and Satisfaction Questionnaire) in which participants respond on a scale of 1 (very poor) to 5 (very good) their level of satisfaction with a variety of social and physical domains. The total raw score ranges from 14 to 70 or 0-100%. Only the first 14 items yield the raw total score as the last two items are standalone. The raw total score is transformed into a percentage maximum possible score using the following formula: (raw total score-minimum score)/(maximum possible raw score-minimum score). The lower values/percentages represent a poor outcome while higher values/percentages represent a better outcome. The information below reflects raw scores (rather than percentages).
Time Frame: Baseline and every 6 months over 2 year active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 426 | 638
Units on a scale
  Baseline | 42.00 (11.60) | 44.38 (11.12)
  6 month follow-up: number analyzed (Participants) | 295 | 499
  6 month follow-up | 42.29 (11.32) | 45.76 (11.09)
  12 month follow-up: number analyzed (Participants) | 250 | 425
  12 month follow-up | 44.52 (10.36) | 44.35 (11.42)
  18 month follow-up: number analyzed (Participants) | 234 | 393
  18 month follow-up | 43.10 (10.75) | 44.88 (11.34)
  24 month follow-up: number analyzed (Participants) | 166 | 355
  24 month follow-up | 43.98 (11.65) | 45.80 (12.02)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.0014, Mixed Models Analysis

7. Secondary Outcome: Change in Medication Adherence - Diabetes
Description: Claims data used to calculate diabetes medication possession ratio (MPO) for participants diagnosed with diabetes in 6 month time periods. If the (first_fill - last_end_Date) > 180 then MPR = (total days supply - (first_fill - last_end_Date) - 180 ) / 180. If the total duration was not greater than 180 days, MPR = total days supply / 180.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: The N for the time point with the greatest # of participants who were prescribed a diabetes medication.
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 47 | 58
Medication possession ratio
  Baseline: number analyzed (Participants) | 40 | 58
  Baseline | 0.78 (0.30) | 0.89 (0.20)
  6 month follow-up: number analyzed (Participants) | 41 | 52
  6 month follow-up | 0.86 (0.27) | 0.91 (0.20)
  12 month follow-up: number analyzed (Participants) | 47 | 55
  12 month follow-up | 0.83 (0.27) | 0.91 (0.17)
  18 month follow-up: number analyzed (Participants) | 35 | 51
  18 month follow-up | 0.86 (0.23) | 0.88 (0.24)
  24 month follow-up: number analyzed (Participants) | 29 | 48
  24 month follow-up | 0.77 (0.32) | 0.91 (0.17)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.0001, Mixed Models Analysis

8. Secondary Outcome: Change in Functional Status (Sheehan Disability Scale)
Description: Functional status is measured using the Sheehan Disability Scale which assesses functional impairment in three domains including: work/school, social and family life. Respondents rate the extent to which work/school, social life and home life or family responsibilities are impaired by symptoms. The three items from the Sheehan Disability Scale are summed together into a single measure of global functional impairment. This measure ranges from 0 to 30, with 0 being unimpaired and 30 being highly impaired.
Time Frame: Baseline and every 6 months over 2 year active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 473 | 686
Units on a scale
  Baseline | 13.82 (9.20) | 12.71 (8.82)
  6 month follow-up: number analyzed (Participants) | 324 | 532
  6 month follow-up | 12.97 (8.87) | 11.33 (8.53)
  12 month follow-up: number analyzed (Participants) | 273 | 466
  12 month follow-up | 12.71 (8.60) | 12.29 (8.62)
  18 month follow-up: number analyzed (Participants) | 251 | 424
  18 month follow-up | 13.58 (8.57) | 12.20 (8.54)
  24 month follow-up: number analyzed (Participants) | 184 | 372
  24 month follow-up | 13.31 (8.69) | 11.90 (8.58)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Treatment by time interaction test; Test type: Superiority; p = 0.5566, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time (only calculated if treatment by time interaction non-significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis

9. Secondary Outcome: Change in Emergent Care Use (Claims Data)
Description: Behavioral and physical health claims data will be obtained to determine frequency of emergent service use for participants over 12-month time periods.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: # of individuals with 80% Medicaid eligibility in the 12 months prior to the data collection time point.
Measure: Mean (Standard Deviation); unit: frequency of visits in 12-month periods
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
frequency of visits in 12-month periods
  Baseline | 3.83 (5.87) | 2.36 (4.32)
  12-month follow up: number analyzed (Participants) | 440 | 620
  12-month follow up | 3.21 (5.07) | 2.37 (4.63)
  24-month follow-up: number analyzed (Participants) | 310 | 582
  24-month follow-up | 2.68 (4.44) | 2.19 (4.08)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.002, Mixed Models Analysis

10. Secondary Outcome: Change in Lab Monitoring - Overall
Description: Frequency of lab tests (glucose, lipids, EKG) in 12 month periods
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: Study participants who were Medicaid eligible for 80% of the year prior to the data collection time point
Measure: Mean (Standard Deviation); unit: frequency of lab tests in 12 mo. period
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
frequency of lab tests in 12 mo. period
  Baseline | 1.67 (2.64) | 1.37 (2.65)
  12 month follow-up: number analyzed (Participants) | 440 | 620
  12 month follow-up | 1.60 (2.79) | 1.49 (2.79)
  24 month follow-up: number analyzed (Participants) | 310 | 582
  24 month follow-up | 1.52 (2.36) | 1.30 (2.70)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.0029, Mixed Models Analysis

11. Secondary Outcome: Change in Patient Satisfaction With Care
Description: Change in patient satisfaction with care was assessed using the Patient Assessment of Care for Chronic Conditions (PACIC). Each item of the PACIC is on a 1 to 5 scale. The total score is the average of all 20 item scores. Higher scores represent increased frequency of structured chronic care.
Time Frame: Baseline and every 6 months over 2 year active intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 444 | 647
Units on a scale
  Baseline | 2.99 (1.06) | 3.17 (0.96)
  6 month follow-up: number analyzed (Participants) | 312 | 522
  6 month follow-up | 3.17 (1.04) | 3.23 (0.95)
  12 month follow-up: number analyzed (Participants) | 260 | 458
  12 month follow-up | 3.25 (0.99) | 3.31 (0.95)
  18 month follow-up: number analyzed (Participants) | 253 | 409
  18 month follow-up | 3.16 (1.03) | 3.25 (0.95)
  24 month follow-up: number analyzed (Participants) | 175 | 358
  24 month follow-up | 3.17 (1.10) | 3.37 (0.95)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.0021, Mixed Models Analysis

12. Secondary Outcome: Change in Medication Adherence - Antipsychotics
Description: Claims data used to calculate antipsychotic medication possession ratio (MPR) for participants in 6 month time periods. If the (first_fill - last_end_Date) > 180 then MPR = (total days supply - (first_fill - last_end_Date) - 180 ) / 180. If the total duration was not greater than 180 days, MPR = total days supply / 180.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: The N for the time point with the greatest # of participants who were prescribed a antipsychotic medication.
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 151 | 198
Medication possession ratio
  Baseline: number analyzed (Participants) | 147 | 198
  Baseline | 0.73 (0.29) | 0.81 (0.26)
  6 month follow-up: number analyzed (Participants) | 151 | 195
  6 month follow-up | 0.70 (0.32) | 0.80 (0.27)
  12 month follow-up: number analyzed (Participants) | 126 | 181
  12 month follow-up | 0.74 (0.32) | 0.82 (0.27)
  18 month follow-up: number analyzed (Participants) | 98 | 156
  18 month follow-up | 0.78 (0.26) | 0.78 (0.28)
  24 month follow-up: number analyzed (Participants) | 73 | 147
  24 month follow-up | 0.78 (0.28) | 0.81 (0.27)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.1183, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time (only calculated if treatment by time interaction non-significant); Test type: Superiority; p = 0.0569, Mixed Models Analysis

13. Secondary Outcome: Change in Medication Adherence - Hypertension
Description: Claims data used to calculate antihypertensive medication possession ratio (MPR) for participants in 6 month time periods. If the (first_fill - last_end_Date) > 180 then MPR = (total days supply - (first_fill - last_end_Date) - 180 ) / 180. If the total duration was not greater than 180 days, MPR = total days supply / 180.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: The N for the time point with the greatest # of participants who were prescribed a antihypertensive medication.
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 98 | 126
Medication possession ratio
  Baseline: number analyzed (Participants) | 92 | 118
  Baseline | 0.75 (0.31) | 0.76 (0.30)
  6 month follow-up | 0.73 (0.31) | 0.79 (0.30)
  12 month follow-up: number analyzed (Participants) | 96 | 125
  12 month follow-up | 0.76 (0.29) | 0.82 (0.27)
  18 month follow-up: number analyzed (Participants) | 86 | 114
  18 month follow-up | 0.81 (0.28) | 0.80 (0.28)
  24 month follow-up: number analyzed (Participants) | 60 | 102
  24 month follow-up | 0.83 (0.30) | 0.82 (0.27)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.0745, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time (only calculated if treatment by time interaction non-significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis

14. Secondary Outcome: Change in Medication Adherence - Antidepressants
Description: Claims data used to calculate antidepressant medication possession ratio (MPR) for participants in 6 month time periods. If the (first_fill - last_end_Date) > 180 then MPR = (total days supply - (first_fill - last_end_Date) - 180 ) / 180. If the total duration was not greater than 180 days, MPR = total days supply / 180.
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: The N for the time point with the greatest # of participants who were prescribed am antidepressant medication.
Measure: Mean (Standard Deviation); unit: Medication possession ratio
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 188 | 231
Medication possession ratio
  Baseline | 0.79 (0.31) | 0.84 (0.27)
  6 month follow-up: number analyzed (Participants) | 176 | 225
  6 month follow-up | 0.79 (0.29) | 0.86 (0.24)
  12 month follow-up: number analyzed (Participants) | 158 | 221
  12 month follow-up | 0.81 (0.27) | 0.84 (0.27)
  18 month follow-up: number analyzed (Participants) | 149 | 202
  18 month follow-up | 0.81 (0.29) | 0.82 (0.27)
  24 month follow-up: number analyzed (Participants) | 102 | 189
  24 month follow-up | 0.83 (0.27) | 0.82 (0.26)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.1653, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time (only calculated if treatment by time interaction non-significant); Test type: Superiority; p = 0.1772, Mixed Models Analysis

15. Secondary Outcome: Change in Lab Monitoring - Glucose
Description: Frequency of glucose lab tests in 12 month periods
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: Study participants who were Medicaid eligible for 80% of the year prior to the data collection time point
Measure: Mean (Standard Deviation); unit: frequency of lab tests in 12 mo. period
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
frequency of lab tests in 12 mo. period
  Baseline | 1.55 (2.55) | 1.21 (2.52)
  12 month follow-up: number analyzed (Participants) | 440 | 620
  12 month follow-up | 1.46 (2.69) | 1.33 (2.65)
  24 month follow-up: number analyzed (Participants) | 310 | 582
  24 month follow-up | 1.41 (2.31) | 1.16 (2.50)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p < 0.0001, Mixed Models Analysis

16. Secondary Outcome: Change in Lab Monitoring - Lipids
Description: Frequency of lipid lab tests in 12 month periods
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: Study participants who were Medicaid eligible for 80% of the year prior to the data collection time point
Measure: Mean (Standard Deviation); unit: frequency of lab tests in 12 mo. period
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
frequency of lab tests in 12 mo. period
  Baseline | 0.37 (0.74) | 0.41 (0.86)
  12 month follow-up: number analyzed (Participants) | 440 | 620
  12 month follow-up | 0.35 (0.73) | 0.46 (0.90)
  24 month follow-up: number analyzed (Participants) | 310 | 582
  24 month follow-up | 0.40 (0.73) | 0.46 (1.39)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.0202, Mixed Models Analysis

17. Secondary Outcome: Change in Lab Monitoring - EKG
Description: Frequency of EKG tests in 12 month periods
Time Frame: Updated annually using claims data over 2 year active intervention period
Population: Study participants who were Medicaid eligible for 80% of the year prior to the data collection time point
Measure: Mean (Standard Deviation); unit: frequency of EKG tests in 12 mo. period
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
Number analyzed (Participants) | 449 | 648
frequency of EKG tests in 12 mo. period
  Baseline | 0.12 (0.39) | 0.15 (0.51)
  12 month follow-up: number analyzed (Participants) | 440 | 620
  12 month follow-up | 0.13 (0.43) | 0.16 (0.49)
  24 month follow-up: number analyzed (Participants) | 310 | 582
  24 month follow-up | 0.10 (0.34) | 0.12 (0.42)
Statistical Analysis 1: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for treatment by time interaction; Test type: Superiority; p = 0.4715, Mixed Models Analysis
Statistical Analysis 2: Comparison: Patient Self-Directed Care vs Provider-Supported Integrated Care; Test for change over time (only calculated if treatment by time interaction non-significant); Test type: Superiority; p = 0.9209, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Over the entire 2 year implementation and data collection period: October 2013 - January 2016
Arm/Group | Patient Self-Directed Care | Provider-Supported Integrated Care
All-Cause Mortality (participants affected / at risk) | 3/516 | 6/713
Serious Adverse Events (participants affected / at risk) | 3/516 | 6/713
Other Adverse Events (participants affected / at risk) | 0/516 | 0/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Self-Directed Care (N=516) | Provider-Supported Integrated Care (N=713)
Death - not associated with study activities (General disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No